CLINICAL TRIAL: NCT05670717
Title: Subsidence of Cementless Stem Following Arthroplasty for Fracture Neck of Femur
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amgad Rasmy Moreed Gerges, principal investigator (resident doctor), Assiut University
Other Study IDs: Subsidence of Cementless Stem
Record Dates: First submitted 2022-05-19; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Hip Arthropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of subsidence of cementless stem following arthroplasty for fracture neck of femur.

DETAILED DESCRIPTION:
Neck of femur fractures are occurring at an increased incidence, Functionally independent patients without cognitive impairment can expect reasonable life expectancy, this indicates the need for a durable surgical option that optimises the chance to return to pre-injury functional status, with minimal risk of complications and reoperation. THA should be considered the gold standard producing better functional and quality of life outcomes lower reoperation rates and better cost effectiveness.

THA is associated with better functional outcomes and a lower risk of revision surgery in self-sufficient, physically active patients , Instability is the leading complication of conventional THA and occurs with a higher incidence ,THA remains the option of choice as it provides better functional outcomes.

Although the clinical outcomes of total hip arthroplasty (THA) in elderly patients with femoral neck fracture were reported to be better than hemiarthroplasty, hemiarthroplasty was frequently recommended in cases where the patient has a low functional level and/or osteoporosis and high rates of postoperative dislocation of total hip arthroplasty.

Hip joint replacement surgery is considered one of the most successful operations due to its high success and low complication rate , one possible risk factor for early failure of total hip arthroplasty (THA) is the subsidence of the femoral stem , Cementless THA in particular could be susceptible to subsidence.

Cementless femoral stems ideally achieve direct integration between the stem surface and endosteal bone with the aim of decreasing the incidence of aseptic loosening.

Subsidence is defined as a distalization of the femoral stem in reference to the greater trochanter.

Measurement of subsidence of uncemented femoral stems can be used to evaluate the likelihood of long term stem component loosening and therefore clinical failure .

ELIGIBILITY:
Inclusion Criteria:

* cases that underwent cementless hip arthroplasty for fracture neck of femur

Exclusion Criteria:

- 1- malignancy. 2- Previous plating. 3- Revision for infection. 4- dysplasia. 5- SLE and Rheumatoid Arthritis

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cases that previously underwent cementless hip arthroplasty for fracture neck of femur at arthroplasty unit at assiut university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of subsidence of cementless stem following arthroplasty for fracture neck of femur. | an average of 1 year post operatively
  Radiological evaluation of stem subsidence by standing anteroposterior radiograph on hip joint 1 year post-operatively to be compared with the previous anteroposterior hip radiograph that was done immediately after operation and assessment of subsidence by measuring the distance between the apex of major trochanter and the stem shoulder or measuring the distance between stem shoulder of hip prosthesis and the most prominent point of lesser trochanter

SECONDARY OUTCOMES:
1- Harris Hip Scoring for assessment pain and distance walked and range of motion and quality of life. 2- Health Survey (SF-36) Scoring.foe assesment of health ststus and daily activities 3- Any complications detected. | 1 year after surgery.

REFERENCES:
- [Background] Guyen O. Hemiarthroplasty or total hip arthroplasty in recent femoral neck fractures? Orthop Traumatol Surg Res. 2019 Feb;105(1S):S95-S101. doi: 10.1016/j.otsr.2018.04.034. Epub 2018 Nov 16. PMID 30449680
- [Background] Burgers PT, Van Geene AR, Van den Bekerom MP, Van Lieshout EM, Blom B, Aleem IS, Bhandari M, Poolman RW. Total hip arthroplasty versus hemiarthroplasty for displaced femoral neck fractures in the healthy elderly: a meta-analysis and systematic review of randomized trials. Int Orthop. 2012 Aug;36(8):1549-60. doi: 10.1007/s00264-012-1569-7. Epub 2012 May 24. PMID 22623062
- [Background] Leiss F, Gotz JS, Meyer M, Maderbacher G, Reinhard J, Parik L, Grifka J, Greimel F. Differences in femoral component subsidence rate after THA using an uncemented collarless femoral stem: full weight-bearing with an enhanced recovery rehabilitation versus partial weight-bearing. Arch Orthop Trauma Surg. 2022 Apr;142(4):673-680. doi: 10.1007/s00402-021-03913-0. Epub 2021 May 21. PMID 34019145
- [Background] Mazoochian F, Schrimpf FM, Kircher J, Mayer W, Hauptmann S, Fottner A, Muller PE, Pellengahr C, Jansson V. Proximal loading of the femur leads to low subsidence rates: first clinical results of the CR-stem. Arch Orthop Trauma Surg. 2007 Aug;127(6):397-401. doi: 10.1007/s00402-007-0384-x. Epub 2007 Jun 30. PMID 17602233
- [Background] Parvizi J, Keisu KS, Hozack WJ, Sharkey PF, Rothman RH. Primary total hip arthroplasty with an uncemented femoral component: a long-term study of the Taperloc stem. J Arthroplasty. 2004 Feb;19(2):151-6. doi: 10.1016/j.arth.2003.10.003. PMID 14973856
- [Background] Ries C, Boese CK, Dietrich F, Miehlke W, Heisel C. Femoral stem subsidence in cementless total hip arthroplasty: a retrospective single-centre study. Int Orthop. 2019 Feb;43(2):307-314. doi: 10.1007/s00264-018-4020-x. Epub 2018 Jun 18. PMID 29916001
- [Background] Al-Najjim M, Khattak U, Sim J, Chambers I. Differences in subsidence rate between alternative designs of a commonly used uncemented femoral stem. J Orthop. 2016 Jul 5;13(4):322-6. doi: 10.1016/j.jor.2016.06.026. eCollection 2016 Dec. PMID 27436922
- [Background] Hoskins W, Webb D, Bingham R, Pirpiris M, Griffin XL. Evidence based management of intracapsular neck of femur fractures. Hip Int. 2017 Sep 19;27(5):415-424. doi: 10.5301/hipint.5000519. Epub 2017 Sep 11. PMID 28956892